CLINICAL TRIAL: NCT07175740
Title: Influence of the Macronutrient Content of a Standardized Pre-Exercise Meal on the Glycemic Response Following Exercise in Type 2 Diabetics
Brief Title: Effect of Macronutrients on Post-Exercise Glycemic Response in Males With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Poirier (Other)
Responsible Party: Sponsor-Investigator, Paul Poirier, Cardiologist, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 859
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Glycemic Response
Keywords: Macronutrients; Type 2 Diabetes; Glycemic response; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Single-blind randomized crossover design with 5 conditions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Fasting (Experimental): Fasting before the exercise intervention
  Interventions: Dietary Supplement: Fasting; Other: Exercise session
- Sucrose (Experimental): Sucrose enriched meal, consumed 2 hours before the exercise intervention
  Interventions: Dietary Supplement: Sucrose enriched meal; Other: Exercise session
- Fructose (Experimental): Fructose meal, consumed 2 hours before the exercise intervention.
  Interventions: Dietary Supplement: Fructose enriched meal; Other: Exercise session
- Aspartame (Experimental): Aspartame enriched meal, consumed 2 hours before the exercise intervention.
  Interventions: Dietary Supplement: Aspartame enriched meal; Other: Exercise session
- Fat (Experimental): Fat enriched meal, consumed 2 hours before the exercise intervention.
  Interventions: Dietary Supplement: Fat enriched meal; Other: Exercise session

INTERVENTIONS:
Dietary Supplement: Fasting — No meal
  Arms: Fasting
Dietary Supplement: Sucrose enriched meal — 175 ml of oatmeal cereal, one slice of bread, 30g of cheese, 22g sucrose
  Arms: Sucrose
Dietary Supplement: Fructose enriched meal — 175 ml of oatmeal cereal, one slice of bread, 30g of cheese, 22g fructose
  Arms: Fructose
Dietary Supplement: Fat enriched meal — 175 ml of oatmeal cereal, one slice of bread, 30g of cheese, 15g fat
  Arms: Fat
Dietary Supplement: Aspartame enriched meal — 175 ml of oatmeal cereal, one slice of bread, 30g of cheese, aspartame (matched for taste)
  Arms: Aspartame
Other: Exercise session — A 60-minutes exercise session on a cycle ergometer (Corival 400, Quinton Instruments, Seattle, WA, USA) at 60% of the VO2peak (determined at a baseline visit)

SUMMARY:
The goal of this randomized crossover trial is to evaluate the impact of meal macronutrient composition on the glycemic response following exercise in males with type 2 diabetes. The main question it aims to answer is:

• Is the consumption of a glucose enriched meal associated with a bigger reduction in plasma glucose following a 1-hour exercise session than other meals Researchers will compare different meal macronutrient composition to see how it affects the glycemic response after exercise.

Participants will

* Fast, then do a 1-hour exercise session
* Eat a glucose enriched meal, then do a 1-hour exercise session
* Eat a fructose enriched meal, then do a 1-hour exercise session
* Eat a fat enriched meal, then do a 1-hour exercise session
* Eat an aspartame enriched meal, then do a 1-hour exercise session

DETAILED DESCRIPTION:
Meals The meals will be equivalent in terms of total calories (with the exception of the aspartame meal) and the percentage of protein will be the same in all four conditions. Only the fat and carbohydrates percentages will vary in the four meal conditions.

Exercise protocol Each subject will perform a maximal aerobic capacity (VO2peak) test on an ergocycle at the start of the protocol. Subsequently, at one-week intervals, each patient will perform an exercise session consisting of one hour of ergocycle at a capacity corresponding to 60% of each individual's VO2peak. The prescribed workload will be established based on the VO2peak test. Exercise will be monitored using heart rate, work, and oxygen consumption measured using an indirect calorimetry system. The five conditions will be randomized and performed at one-week intervals. Each exercise session will be supervised by a physician. Patients taking oral hypoglycemic agents will not take their medication on the morning of the exercise.

Blood samples Samples will be taken to measure glucose, free fatty acids, insulin, glucagon, and plasma catecholamines. In addition, an indirect calorimetry system will allow us to measure total substrate oxidation. For each blood sample period, there will be a 5-minute assessment as described above.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Oral hypoglycemic agents

Exclusion Criteria:

* Insulin
* Other diabetes related medical complications or conditions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-05-30 (Actual); Primary Completion 2004-05-28 (Actual); Study Completion 2004-05-28 (Actual)

PRIMARY OUTCOMES:
Glycemic response during and following intervention | Plasma glucose and insulin levels from blood samples taken at -15, 0, 15, 30, 45, 60, 75 and 90 minutes from the beginning of the exercise.
  Plasma glucose and insulin levels following consumption of different meal compositions and following a 1-hour exercise session.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada